CLINICAL TRIAL: NCT00712114
Title: A Phase I/II, Open Label, Dose Ranging Study of the Safety, Tolerance, Pharmacokinetics and Potential Anti-Inflammatory Activity of HE3286 When Administered Orally for 29 Days to Patients With Rheumatoid Arthritis on a Stable Dose of Methotrexate
Brief Title: Safety, Tolerance, Pharmacokinetics and Activity of HE3286 in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Harbor Therapeutics (Industry)
Responsible Party: Nanette Onizuka-Handa/Sr. Vice President, Regulatory Affairs and Quality, Hollis-Eden Pharmaceuticals
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE3286-0201
Record Dates: First submitted 2008-07-06; First posted 2008-07-09 (Estimated); Last update posted 2011-06-14 (Estimated); Status verified 2011-06

CONDITIONS: Rheumatoid Arthritis
Keywords: phase I; safety; tolerance; rheumatoid arthritis; pharmacokinetics; methotrexate; anti-inflammatory
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — 17-ethynyl-5-androstene-3, 7, 17-triol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 (Experimental): 10 mg HE3286 (1 x 5 mg HE3286, BID)
  Interventions: Drug: HE3286
- Cohort 2 (Experimental): 20 mg HE3286 (2 x 5 mg HE3286 BID)
  Interventions: Drug: HE3286
- Cohort 3 (Experimental): 40 mg HE3286 (4 x 5 mg HE3286 BID)
  Interventions: Drug: HE3286

INTERVENTIONS:
Drug: HE3286 — HE3286 will be administered orally. Dosing will be 10 mg per day for 29 days.
  Other Names: Triolex
  Arms: Cohort 1
Drug: HE3286 — HE3286 will be administered orally. Dosing will be 20 mg per day for 29 days
  Other Names: Triolex
  Arms: Cohort 2
Drug: HE3286 — HE3286 will be administered orally. Dosing will be 40 mg per day for 29 days
  Other Names: Triolex
  Arms: Cohort 3

SUMMARY:
The purpose of this pilot, exploratory study is to evaluate the safety, tolerance, pharmacokinetics and potential anti-inflammatory activity of an investigational agent, HE3286, when administered orally for 29 days to patients with rheumatoid arthritis that are taking a stable dose of methotrexate.

DETAILED DESCRIPTION:
This is a Phase I/II, open label, dose ranging study of the safety, tolerance, and anti-inflammatory activity of HE3286 in patients with rheumatoid arthritis. Patients will receive study treatment (one of three open label doses) in addition to their current stable dose of methotrexate. Safety (via monitoring of vital signs, physical examination changes, ECG results, laboratory results, and adverse events), pharmacokinetics profiles (of HE3286 and methotrexate) and anti-inflammatory activity will be assessed over a treatment period of 29 days.

ELIGIBILITY:
Main Inclusion Criteria:

* Male or female patient 18-75 years of age
* Patient with stable or active disease on a stable dose of methotrexate for at least 30 days prior to Day 1
* Patient has normal thyroid stimulating hormone (TSH) levels with or without thyroid replacement therapy
* Patient is willing to abstain from consuming grapefruit containing products from 24 hours prior to dosing until the end of the study as it may affect the pharmacokinetic measurements
* Patient has not experienced renal or liver disease by history and/or based on laboratory results
* Patient has not experienced acute cardiac disease within 6 months prior to Screening
* Patient must provide voluntary, written, informed consent prior to screening evaluations and be able to follow verbal and written instructions.

Main Exclusion Criteria:

* Functional status class IV according to The American College of Rheumatology (ACR) criteria
* Patient who has a history of clinically significant cardiovascular disease (including coronary artery disease), clinically significant hepatic, respiratory or renal abnormalities, or clinically significant endocrine disorders (including diabetes)
* Patient with active Tuberculosis (TB) or evidence of latent TB without previous adequate therapy
* Systemic autoimmune disorder (including, but not limited to, systemic lupus erythematosus, inflammatory bowel disease, scleroderma, inflammatory myopathy, mixed connective tissue disease or any overlap syndrome)
* Inflammatory joint disease other than RA
* Patient who has received any of the following immunosuppressive drugs:

  * Etanercept within 1 month of Day 1;
  * Abatacept, adalimumab, infliximab, leflunomide, imuran, cyclosporin, anakinra, sulfasalazine, bextra, celebrex or gold within 2 months of Day 1 or for biological agents 6 half lives, whichever is greater;
  * Rituximab within 1 year of Day 1
* Patient that is bed or wheelchair bound
* Patients taking prednisone within 2 weeks prior to Screening
* Patient requiring or receiving any of the following within thirty (30) days prior to the screening visit: interleukins, steroids (i.e., anabolic steroids, glucocorticoids), hormone replacement therapy (except stable low-dose HRT for at least 6-months prior to screening), birth control pills, anti-cancer chemotherapeutic agents (except methotrexate), metabolic inhibitors (except methotrexate), concomitant medications that prolong the QT/QTc interval
* Patient who has any clinically significant abnormalities in laboratory results at Screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-07; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Safety and pharmacokinetics | Duration of the study

SECONDARY OUTCOMES:
To assess the potential activity of HE3286 to decrease inflammation via evaluation of inflammatory cytokine activity. | Duration of study

CONTACTS AND LOCATIONS:
Overall Officials: Dwight Stickney, MD, Study Director — Hollis-Eden
Locations (1):
- Beverly Hills, California, United States